CLINICAL TRIAL: NCT00554528
Title: Arthroplasty Versus Fusion in Anterior Cervical Surgery: Prospective Study of the Impact on the Adjacent Level
Acronym: PROCERV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 06-APN-01
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Clinical Radiculopathy; Myelopathy Due to a Cervical Disk Disease
Keywords: Cervical; disc; prosthesis; adjacent; disease; randomized; prospective; study
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): patient receiving cervical disc prosthesis with a mobile insert named Mobi-C and product by LDR médical
  Interventions: Device: cervical disc prosthesis with a mobile insert named Mobi-C
- B (Other): patient receiving intersomatic cage
  Interventions: Procedure: arthrodesis - cervical disk surgery

INTERVENTIONS:
Device: cervical disc prosthesis with a mobile insert named Mobi-C — Stage 1: partial discectomy
  stage 2: location of the medial axis
  stage 3: centering pin
  stage 4: installation of the caspar spacer
  stage 5: total discectomy
  stage 6: parallel distraction
  stage 7: depth measurement
  stage 8: trial implant
  stage 9: assembly
  stage 10: implant insertion
  stage 11: anchorage optimization
  Arms: A
Procedure: arthrodesis - cervical disk surgery — discectomy and arthrodesis
  Arms: B

SUMMARY:
The aim of the study is to evaluate the impact of the cervical disk surgery on the deterioration of the adjacent levels. The investigators compare the radiological deterioration of adjacent levels, at 3 years, in both situation of fusion and arthroplasty. 220 patients are enrolled and randomized to receive fusion or prosthesis. Radiological and clinical follow-up is organized for a period of 3 years.

DETAILED DESCRIPTION:
Anterior surgery of the cervical spine is one of the most practiced procedures in spine surgery. Its immediate accuracy and safety is proved since a long time in case of degenerative disk disease or disk herniation. But the segmental arthrodesis leads to an overload of the adjacent disk. A lot of studies have shown that the increasing mobility and pressure of the adjacent segments can be responsible of new degeneration and clinical symptoms. Recently, cervical disk prosthesis have been developed to maintain the mobility at the level of the surgery. This technique is supposed to decrease the risk of adjacent disk disease but, at this time, the analysis of the results is difficult, due to the lack of randomized studies with long term follow up.

The aim of our prospective randomized study is to evaluate the aftermath of the arthroplasty compared to the fusion on the adjacent disk degeneration.

The main objective is to show a radiological difference at 3 years in term of adjacent disk degeneration.

The secondary objectives are:

* evaluate the rate of new clinical symptoms during three years
* show differences during the postoperative period, especially concerning the length of the hospital stay, the use of pain killers and return to work.
* verify the maintaining of mobility pf the prosthesis during three years.

This is a controlled study with two group of equal size: one group is treated by discectomy and arthrodesis and the other by discectomy and prosthesis/ The criteria for the inclusion of the patients are: clinical radiculopathy and/or myelopathy due to a cervical disk disease (disk herniation or osteophytosis), lack of effect of the medical treatment, CT scan or MRI showing a compression of roots and/or spinal cord.

The main exclusion criteria are: plurisegmental disk disease, injuries happened during professional activities, previous cervical surgery.

During the study, we perform a clinical (standardized scales: Neck Disability Index, Short Form 36, and neurological exam) and a radiological (height of the adjacent disks, ostheophytis,…) follow-up.

The analysis of the current literature and statistical process leads to a total amount of 220 patients enrolled in the study. This is a multicentric study organized for a total duration of five years (two years for inclusions and three years of follow-up).

ELIGIBILITY:
Inclusion Criteria:

* clinical radiculopathy
* myelopathy due to a cervical disk disease
* lack of effect of the medical treatment
* CT scan or MRI showing a compression of roots and/or spinal cord

Exclusion Criteria:

* plurisegmenta disk disease
* injuries happened during professional activities
* previous cervical surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2007-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
show significant difference of degeneration of disc above and below the operated stage between the two groups | 3 years after surgery

SECONDARY OUTCOMES:
show difference of neurological pain between the two groups | during the 3 years of follow-up
show difference of duration of hospitalization and consumption of medication | during the first month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephane LITRICO, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Department of Neurosurgery, CHU de Nice, Nice, France

REFERENCES:
- [Background] Dmitriev AE, Cunningham BW, Hu N, Sell G, Vigna F, McAfee PC. Adjacent level intradiscal pressure and segmental kinematics following a cervical total disc arthroplasty: an in vitro human cadaveric model. Spine (Phila Pa 1976). 2005 May 15;30(10):1165-72. doi: 10.1097/01.brs.0000162441.23824.95. PMID 15897831
- [Background] Eck JC, Humphreys SC, Lim TH, Jeong ST, Kim JG, Hodges SD, An HS. Biomechanical study on the effect of cervical spine fusion on adjacent-level intradiscal pressure and segmental motion. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2431-4. doi: 10.1097/00007632-200211150-00003. PMID 12435970
- [Background] Hilibrand AS, Robbins M. Adjacent segment degeneration and adjacent segment disease: the consequences of spinal fusion? Spine J. 2004 Nov-Dec;4(6 Suppl):190S-194S. doi: 10.1016/j.spinee.2004.07.007. PMID 15541666
- [Background] Goffin J, Geusens E, Vantomme N, Quintens E, Waerzeggers Y, Depreitere B, Van Calenbergh F, van Loon J. Long-term follow-up after interbody fusion of the cervical spine. J Spinal Disord Tech. 2004 Apr;17(2):79-85. doi: 10.1097/00024720-200404000-00001. PMID 15260088
- [Background] Link HD, McAfee PC, Pimenta L. Choosing a cervical disc replacement. Spine J. 2004 Nov-Dec;4(6 Suppl):294S-302S. doi: 10.1016/j.spinee.2004.07.022. PMID 15541680
- [Background] Albert TJ, Eichenbaum MD. Goals of cervical disc replacement. Spine J. 2004 Nov-Dec;4(6 Suppl):292S-293S. doi: 10.1016/j.spinee.2004.07.023. PMID 15541679
- [Background] McAfee PC. The indications for lumbar and cervical disc replacement. Spine J. 2004 Nov-Dec;4(6 Suppl):177S-181S. doi: 10.1016/j.spinee.2004.07.003. PMID 15541664
- [Background] Fager CA. Cervical arthroplasty. J Neurosurg Spine. 2005 Mar;2(3):394-5; author reply 395. doi: 10.3171/spi.2005.2.3.0394. No abstract available. PMID 15796370
- [Background] Phillips FM, Garfin SR. Cervical disc replacement. Spine (Phila Pa 1976). 2005 Sep 1;30(17 Suppl):S27-33. doi: 10.1097/01.brs.0000175192.55139.69. PMID 16138062
- [Background] Pracyk JB, Traynelis VC. Treatment of the painful motion segment: cervical arthroplasty. Spine (Phila Pa 1976). 2005 Aug 15;30(16 Suppl):S23-32. doi: 10.1097/01.brs.0000174507.45083.98. PMID 16103831
- [Background] Hacker RJ. Cervical disc arthroplasty: a controlled randomized prospective study with intermediate follow-up results. Invited submission from the joint section meeting on disorders of the spine and peripheral nerves, March 2005. J Neurosurg Spine. 2005 Dec;3(6):424-8. doi: 10.3171/spi.2005.3.6.0424. PMID 16381203
- [Background] Robertson JT, Papadopoulos SM, Traynelis VC. Assessment of adjacent-segment disease in patients treated with cervical fusion or arthroplasty: a prospective 2-year study. J Neurosurg Spine. 2005 Dec;3(6):417-23. doi: 10.3171/spi.2005.3.6.0417. PMID 16381202
- [Background] Singh M, Gopinath R. Topical analgesia for chest tube removal in cardiac patients. J Cardiothorac Vasc Anesth. 2005 Dec;19(6):719-22. doi: 10.1053/j.jvca.2005.07.024. PMID 16326294
- [Background] Chi JH, Ames CP, Tay B. General considerations for cervical arthroplasty with technique for ProDisc-C. Neurosurg Clin N Am. 2005 Oct;16(4):609-19, vi. doi: 10.1016/j.nec.2005.07.001. PMID 16326284
- [Background] Bertagnoli R, Yue JJ, Pfeiffer F, Fenk-Mayer A, Lawrence JP, Kershaw T, Nanieva R. Early results after ProDisc-C cervical disc replacement. J Neurosurg Spine. 2005 Apr;2(4):403-10. doi: 10.3171/spi.2005.2.4.0403. PMID 15871478
- [Background] Puttlitz CM, Rousseau MA, Xu Z, Hu S, Tay BK, Lotz JC. Intervertebral disc replacement maintains cervical spine kinetics. Spine (Phila Pa 1976). 2004 Dec 15;29(24):2809-14. doi: 10.1097/01.brs.0000147739.42354.a9. PMID 15599283
- [Background] Puttlitz CM, DiAngelo DJ. Cervical spine arthroplasty biomechanics. Neurosurg Clin N Am. 2005 Oct;16(4):589-94, v. doi: 10.1016/j.nec.2005.07.002. PMID 16326281
- [Background] Pickett GE, Rouleau JP, Duggal N. Kinematic analysis of the cervical spine following implantation of an artificial cervical disc. Spine (Phila Pa 1976). 2005 Sep 1;30(17):1949-54. doi: 10.1097/01.brs.0000176320.82079.ce. PMID 16135984
- [Background] Parkinson JF, Sekhon LH. Cervical arthroplasty complicated by delayed spontaneous fusion. Case report. J Neurosurg Spine. 2005 Mar;2(3):377-80. doi: 10.3171/spi.2005.2.3.0377. PMID 15796366
- [Background] Murray BE, Lopardo HA, Rubeglio EA, Frosolono M, Singh KV. Intrahospital spread of a single gentamicin-resistant, beta-lactamase-producing strain of Enterococcus faecalis in Argentina. Antimicrob Agents Chemother. 1992 Jan;36(1):230-2. doi: 10.1128/AAC.36.1.230. PMID 1590694
- [Background] Bertagnoli R, Duggal N, Pickett GE, Wigfield CC, Gill SS, Karg A, Voigt S. Cervical total disc replacement, part two: clinical results. Orthop Clin North Am. 2005 Jul;36(3):355-62. doi: 10.1016/j.ocl.2005.02.009. PMID 15950695
- [Background] Pickett GE, Sekhon LH, Sears WR, Duggal N. Complications with cervical arthroplasty. J Neurosurg Spine. 2006 Feb;4(2):98-105. doi: 10.3171/spi.2006.4.2.98. PMID 16506475